CLINICAL TRIAL: NCT04264533
Title: Vitamin C Infusion for the Treatment of Severe 2019-nCoV Infected Pneumonia: a Prospective Randomized Clinical Trial
Brief Title: Vitamin C Infusion for the Treatment of Severe 2019-nCoV Infected Pneumonia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: the study was started in the second half of the outbreak, and the number of qualifying COVID-19 patients decreased with the control of the epidemic so that we had to stop our trial before reaching the predefined sample size.
Sponsor: ZhiYong Peng (Other)
Responsible Party: Sponsor-Investigator, ZhiYong Peng, Professor; Chief physician, Zhongnan Hospital
Organization: Zhongnan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020001
Record Dates: First submitted 2020-02-04; First posted 2020-02-11 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Vitamin C; Pneumonia, Viral; Pneumonia, Ventilator-Associated
Keywords: Vitamin C; 2019-novel coronavirus pneumonia; Severe acute respiratory infection
MeSH Terms: conditions — Pneumonia, Viral; Pneumonia, Ventilator-Associated | interventions — Ascorbic Acid; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VC (Experimental): 12g Vitamin C+sterile water for injection; total volume: 50ml. 12ml/h; infusion pump；q12h.
  Interventions: Drug: VC
- Sterile water for injection (Placebo Comparator): 50ml water for injection. 12ml/h; infusion pump; q12h.
  Interventions: Drug: Sterile Water for Injection

INTERVENTIONS:
Drug: VC — 12g Vitamin C will be infused in the experimental group twice a day for 7 days by the infusion pump with a speed of 12ml/h.
  Other Names: Vitamin C
  Arms: VC
Drug: Sterile Water for Injection — 50ml sterile water for injection will be infused in the placebo comparator group twice a day for 7 days by the infusion pump with a speed of 12ml/h.
  Arms: Sterile water for injection

SUMMARY:
2019 new coronavirus (2019-nCoV) infected pneumonia, namely severe acute respiratory infection (SARI) has caused global concern and emergency. There is a lack of effective targeted antiviral drugs, and symptomatic supportive treatment is still the current main treatment for SARI.

Vitamin C is significant to human body and plays a role in reducing inflammatory response and preventing common cold. In addtion, a few studies have shown that vitamin C deficiency is related to the increased risk and severity of influenza infections.

We hypothize that Vitamin C infusion can help improve the prognosis of patients with SARI. Therefore, it is necessary to study the clinical efficacy and safety of vitamin C for the clinical management of SARI through randomized controlled trials during the current epidemic of SARI.

DETAILED DESCRIPTION:
At the end of 2019, patients with unexplained pneumonia appeared in Wuhan, China. At 21:00 on January 7, 2020, a new coronavirus was detected in the laboratory, and the detection of pathogenic nucleic acids was completed at 20:00 on January 10. Subsequently, the World Health Organization officially named the new coronavirus that caused the pneumonia epidemic in Wuhan as 2019 new coronavirus (2019-nCoV), and the pneumonia was named severe acute respiratory infection (SARI). Up to February 4, 2020, over 20000 cases have been diagnosed in China, 406 of which have died, and 154 cases have been discovered in other countries around the world. Most of the deaths were elderly patients or patients with severe underlying diseases. SARI has caused global concern and emergency.

Statistics of the 41 patients with SARI published in JAMA initially showed that 13 patients were transferred into the ICU, of which 11 (85%) had ARDS and 3 (23%) had shock. Of these, 10 (77%) required mechanical ventilation support, and 2 (15%) required ECMO support. Of the above 13 patients, 5 (38%) eventually died and 7 (38%) were transferred out of the ICU. Viral pneumonia is a dangerous condition with a poor clinical prognosis. For most viral infections, there is a lack of effective targeted antiviral drugs, and symptomatic supportive treatment is still the current main treatment.

Vitamin C, also known as ascorbic acid, has antioxidant properties. When sepsis happens, the cytokine surge caused by sepsis is activated, and neutrophils in the lungs accumulate in the lungs, destroying alveolar capillaries. Early clinical studies have shown that vitamin C can effectively prevent this process. In addition, vitamin C can help to eliminate alveolar fluid by preventing the activation and accumulation of neutrophils, and reducing alveolar epithelial water channel damage. At the same time, vitamin C can prevent the formation of neutrophil extracellular traps, which is a biological event of vascular injury caused by neutrophil activation. Vitamins can effectively shorten the duration of the common cold. In extreme conditions (athletes, skiers, art workers, military exercises), it can effectively prevent the common cold. And whether vitamin C also has a certain protective effect on influenza patients, only few studies have shown that vitamin C deficiency is related to the increased risk and severity of influenza infections. In a controlled but non-randomized trial, 85% of the 252 students treated experienced a reduction in symptoms in the high-dose vitamin C group (1g / h at the beginning of symptoms for 6h, followed by 3 * 1g / day). Among patients with sepsis and ARDS, patients in the high-dose vitamin group did not show a better prognosis and other clinical outcomes. There are still some confounding factors in the existing research, and the conclusions are different.

Therefore, during the current epidemic of SARI, it is necessary to study the clinical efficacy and safety of vitamin C for viral pneumonia through randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old;
2. Diagnosed as serious or critical SARI (according to the 4th version of Diagnosis and Clinical management of 2019-nCoV infected pneumonia);
3. Being treated in the ICU.

Exclusion Criteria:

1. Allergic to vitamin C;
2. Dyspnea due to cardiogenic pulmonary edema;
3. Pregnant or breastfeeding;
4. Expected life is less than 24 hours;
5. There is a state of tracheotomy or home oxygen therapy in the past;
6. Previously complicated with end-stage lung disease, end-stage malignancy, glucose-6-phosphate dehydrogenase deficiency, diabetic ketoacidosis, and active kidney stone disease;
7. The patient participates in another clinical trial at the same time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-29 (Actual)

PRIMARY OUTCOMES:
Ventilation-free days | on the day 28 after enrollment
  days without ventilation support during 28 days after patients' enrollment

SECONDARY OUTCOMES:
28-days mortality | on the day 28 after enrollment
  wether the patient survives
ICU length of stay | on the day 28 after enrollment
  days of the patients staying in the ICU
Demand for first aid measuments | on the day 28 after enrollment
  the rate of CPR
Vasopressor days | on the day 28 after enrollment
  days of using vasopressors
Respiratory indexes | on the day 10 and 28 after enrollment
  P O2/Fi O2 which reflects patients' respiratory function
Ventilator parameters | on the day 10 and 28 after enrollment
  Ecmo or ventilator
APACHE II scores | on the day 10 after enrollment
  Acute Physiology and Chronic Health Evaluation
SOFA scores | on the day 10 after enrollment
  Sepsis-related Organ Failure Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyong Peng, professor, Principal Investigator — Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu F, Zhu Y, Zhang J, Li Y, Peng Z. Intravenous high-dose vitamin C for the treatment of severe COVID-19: study protocol for a multicentre randomised controlled trial. BMJ Open. 2020 Jul 8;10(7):e039519. doi: 10.1136/bmjopen-2020-039519. PMID 32641343